CLINICAL TRIAL: NCT05870098
Title: Meatal Swab Yourself With Testing for Infections Collectively (MYSTIC)
Brief Title: Meatal Swab Yourself With Testing for Infections Collectively
Acronym: MYSTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GU19-125925
Record Dates: First submitted 2023-04-28; First posted 2023-05-23 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Chlamydia; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Intervention Model Description: Diagnostic accuracy study Single group receiving standard care plus two new comparators
Masking Description: Laboratory staff will be masked and will not be able to link pooled samples (sent under a unique study number) to comparator standard care separate samples (sent under a unique patient identifier).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants will receive:
  1. Clinician or self-taken, pharyngeal and rectal swabs with FCU analysed individually
  2. Self-taken pharyngeal, meatal, and rectal swabs analysed as a pooled specimen
  3. Self-taken pharyngeal and rectal swabs with 1.5ml FCU analysed as a pooled specimen The FCU will be done after any meatal swabs. Patients will be instructed to only pass the first 5ml into the tube, and the tube will be pre-marked with a black line. Full pictoral instructions and verbal support will be given to enable them to complete the pooling process of the swabs and urine.
  Interventions: Diagnostic Test: All participants

INTERVENTIONS:
Diagnostic Test: All participants — 1. Clinician or self-taken, pharyngeal and rectal swabs with FCU analysed individually
  2. Self-taken pharyngeal, meatal, and rectal swabs analysed as a pooled specimen
  3. Self-taken pharyngeal and rectal swabs with 1.5ml FCU analysed as a pooled specimen The FCU will be done after any meatal swabs. Patients will be instructed to only pass the first 5ml into the tube, and the tube will be pre-marked with a black line. Full pictoral instructions and verbal support will be given to enable them to complete the pooling process of the swabs and urine.

SUMMARY:
The goal of this study is

1. to improve the accuracy of chlamydia multi-site testing in men who have sex with men (MSM) and trans-women, whilst saving diagnostic costs, by comparing two new pooling methods with the 3-samples tested separately
2. to assess the diagnostic accuracy of pooled specimens for lymphogranuloma venereum detection (LGV) - a type of chlamydia infection

Chlamydia and gonorrhoea testing for MSM and trans-women usually involves 3 samples from the throat, bum and wee-pipe. The tests can be combined into a single sample pot (pooled sample) which reduces costs, but in a previous study this reduced the accuracy for finding chlamydia.

The main question for this study is:

Can the accuracy of chlamydia testing in a pooled sample be improved by reducing the amount of urine added to minimise dilution, or by using a meatal sample instead of a urine sample?

Participants will be asked to complete two sets of their own throat and bum samples, and then combine these into two pooled samples with 1)a meatal swab and 2)a smaller amount of first catch urine. The order of these samples will be randomised. These samples will be compared against separate samples taken at the same visit, to see how accurate the pooled samples are at diagnosing chlamydia and gonorrhoea with the different sampling techniques.

DETAILED DESCRIPTION:
Testing for chlamydia and gonorrhoea in men who have sex with men (MSM) and trans-women is recommended every three months for those taking HIV Pre-Exposure Prophylaxis (PrEP). Testing requires throat and bottom samples, and samples from the urethra (wee-pipe), usually a urine sample. However, many sexual health services struggle to afford the costs of these 3-samples, four-times per year, which may restrict numbers given PrEP.

The investigators' previous research has shown that the 3-samples (throat, bottom, urine) can be combined into one pooled specimen to accurately find gonorrhoea and reduce laboratory costs. However, the chlamydia results of pooled samples were not as good, finding only 92 out of 100 infections compared with 99 out of 100 with 3 separate samples. The investigators' past research showed no difference in diagnostic accuracy between clinician and self-taken rectum and pharynx swabs for NG and CT detection. People prefer to take their own swabs and self-taken swabs were more cost effective than clinician taken. Self-taken swabs are now used routinely in clinical practice and are available as on-line ordered commercial kits.

This study aims to improve the accuracy of chlamydia results by comparing two new pooling methods with the 3-samples tested separately.

MSM, and trans-women, aged 18 years or over, attending a large UK city sexual health service for chlamydia and gonorrhoea testing will be invited to take part in the study.

The pooling methods will be: 1) pooling with a smaller amount of urine to reduce the dilution of the other samples; and 2) pooling with a swab sample from the outside of the tip of the penis (meatal swab) instead of urine. Meatal swabs are taken by the person themselves. The swab does not go inside the penis so is easy to do and not painful. Studies suggest meatal swabs may be better at finding chlamydia than urine samples.

To ensure an accurate comparison, the order of taking the two pooling method samples, and the 3-samples tested separately, will be randomised.

The study will recruit 1250 participants. This is a large enough number to show if either of the pooling methods can detect more chlamydia than 92 out of 100 infections.

If a pooling technique was developed for MSM and trans-women that did not reduce diagnostic sensitivity, this would likely be implemented. A sensitive, low-cost, method of triple-site STI testing, available on-line, or using minimal in-house staff, would enable increased testing. The investigators believe this study will identify such a method by using meatal swabs or a reduced urine volume. The reduced diagnostic costs of almost two-thirds would enable sexual health clinics to provide PrEP to more people, and/or utilise the money saved elsewhere in their service.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over. Willing to perform self-taken swabs in addition to any clinician required swabs. Able to provide informed consent

Exclusion Criteria:

- Antibiotics taken in the past 14 days (excluding metronidazole). Previous participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males who have sex with males, and trans-females with a penis
Enrollment: 1250 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-05-29 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity for gonorrhoea, chlamydia and LGV diagnosis using NAATS | 14 months
  To improve the accuracy of chlamydia diagnoses in MSM and trans-women by comparing two new pooling methods with the 3-samples tested separately, and to assess the diagnostic accuracy of pooled specimens for lymphogranuloma venereum detection (LGV) - a type of chlamydia infection

SECONDARY OUTCOMES:
Participant satisfaction with using meatal swabs compared with first catch urine for the diagnosis of gonorrhoea, chlamydia, and LGV as measured by a Likert scale | 14 months
  To assess participant satisfaction with using self-taken meatal swabs compared with FCU, participants will complete a questionnaire following their self sampling. Satisfaction will be assessed using a 5 point Likert scale, checking for ease of use, discomfort when sampling, and belief in validity of results.
Participant satisfaction with taking and pooling combined site samples, compared with individually analysed samples for the diagnosis of gonorrhoea, chlamydia, and LGV as measured by a Likert scale | 14 months
  To assess participant satisfaction with taking and pooling combined site samples compared with individually analysed samples, participants will complete a questionnaire following their self sampling. Satisfaction will be assessed using a 5 point Likert scale, checking for ease of process, clarity of instructions, and belief in validity of results.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wilson, MB ChB, Principal Investigator — Leeds Teaching Hospitals NHS Trust; Harriet Wallace, MB ChB, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No